CLINICAL TRIAL: NCT03935074
Title: Superselective Intra-arterial Chemotherapy Treatment for Retinoblastoma- 5 Year Results From Turkey
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Bilge Batu Oto, Ophthalmology Specialist, Medical Doctor, Istanbul University - Cerrahpasa
Other Study IDs: 10136532
Record Dates: First submitted 2019-04-30; First posted 2019-05-02 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Retinoblastoma
Keywords: enucleation; globe salvage; superselective intra-arterial chemotherapy
MeSH Terms: conditions — Retinoblastoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- group 1: Patients who received intra-arterial chemotherapy as a first line treatment
  Interventions: Drug: intra-arterial administration of melphalan
- group 2: Patients who received intra-arterial chemotherapy as a salvage treatment after systemic chemotherapy
  Interventions: Drug: intra-arterial administration of melphalan

INTERVENTIONS:
Drug: intra-arterial administration of melphalan

SUMMARY:
Retrospective review of 5-year long term outcomes of superselective intra-arterial chemotherapy treatment in retinoblastoma in a single institute.

The treatment outcomes, globe salvage rates and complications of superselective intra-arterial chemotherapy both for treating naive patients (primary treatment group) and for patients who received systemic chemotherapy previously (secondary treatment group) were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with unilateral/bilateral retinoblastoma

Exclusion Criteria:

* patients with trilateral retinoblastoma
* extraoculer involvement
* patients with blood dyscrasias, bleeding and clotting disorders

Ages: 5 Months to 7 Years | Sex: All
Age Groups: Child
Study Population: Patients diagnosed with retinoblastoma and who received superselective intra-arterial chemotherapy as a first line treatment or as a salvage treatment after systemic chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-08-30 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
globe salvage | 2-5 years
  globe salvage rate after superselective intra-arterial chemotherapy treatment for retinoblastoma

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University Cerrahpasa School of Medicine Ophthalmology Department, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saglam M, Sarici A, Anagnostakou V, Yildiz B, Kocer N, Islak C, Kizilkilic O. An alternative technique of the superselective catheterization of the ophthalmic artery for intra-arterial chemotherapy of the retinoblastoma: retrograde approach through the posterior communicating artery to the ophthalmic artery. Neuroradiology. 2014 Sep;56(9):751-4. doi: 10.1007/s00234-014-1388-1. Epub 2014 Jun 10. PMID 24913287